CLINICAL TRIAL: NCT04332991
Title: Outcomes Related to COVID-19 Treated With Hydroxychloroquine Among In-patients With Symptomatic Disease
Acronym: ORCHID
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Boyd Taylor Thompson, Co-Prinicipal Investigator PETAL CCC, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PETAL 05 Orchid
Record Dates: First submitted 2020-03-31; First posted 2020-04-03 (Actual); Results first posted 2021-03-17 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Coronavirus; Acute Respiratory Infection; SARS-CoV Infection
Keywords: COVID-19
MeSH Terms: conditions — Coronavirus Infections; Severe Acute Respiratory Syndrome; COVID-19 | interventions — Hydroxychloroquine

STUDY DESIGN:
Intervention Model Description: Eligible participants will be randomized 1:1 to hydroxychloroquine versus placebo. Randomization will be stratified by site and be in permuted blocks of variable size.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients, treating clinicians, trial personnel, and outcome assessors will be blinded to group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Hydroxychlorquine (Active Comparator): Participants assigned to the hydroxychloroquine arm will receive hydroxychloroquine sulfate 400 mg twice daily on the day of enrollment, then 200 mg twice daily for the next 4 days for a 5 day total course.
  Interventions: Drug: Hydroxychloroquine
- Placebo (Placebo Comparator): Participants randomized to the control group will receive a dose of placebo enterally twice daily for 5 days (a total of 10 doses). The placebo pills will be as similar as possible to the hydroxychloroquine pills to ensure blinding.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hydroxychloroquine — Hydroxychloroquine is available in 200 mg oral tablets of hydroxychloroquine sulfate.
  For this COVID-19 trial, we will use an oral or enteral dose of hydroxychloroquine 400 mg twice daily on the day of enrollment, then 200 mg twice daily for the next 4 days for a 5 day total course.
  Arms: Hydroxychlorquine
Drug: Placebo — Participants randomized to the control group will receive a dose of placebo enterally twice daily for 5 days (a total of 10 doses). The placebo pills will be as similar as possible to the hydroxychloroquine pills to ensure blinding.
  Arms: Placebo

SUMMARY:
ORCHID is a multicenter, blinded, placebo-controlled, randomized clinical trial evaluating hydroxychloroquine for the treatment of adults hospitalized with COVID-19. Patients, treating clinicians, and study personnel will all be blinded to study group assignment.

DETAILED DESCRIPTION:
Effective therapies for COVID-19 are urgently needed. Hydroxychloroquine is an antimicrobial agent with immunomodulatory and antiviral properties that has demonstrated in vitro activity against SARS-CoV-2, the virus that causes COVID-19. Preliminary reports suggest potential efficacy in small human studies. Clinical trial data are needed to determine whether hydroxychloroquine is effective in treating COVID-19.

Study Aim: To compare the effect of hydroxychloroquine versus placebo on clinical outcomes, measured using the COVID Ordinal Outcomes Scale at Day 15, among adults with COVID-19 requiring hospitalization.

Study Hypothesis: Among adults hospitalized with COVID-19, administration of hydroxychloroquine will improve clinical outcomes at Day 15.

.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Currently hospitalized or in an emergency department with anticipated hospitalization.
3. Symptoms of acute respiratory infection, defined as one or more of the following:

   1. cough
   2. fever (> 37.5° C / 99.5° F)
   3. shortness of breath (operationalized as any of the following: subjective shortness of breath reported by patient or surrogate; tachypnea with respiratory rate ≥22 /minute; hypoxemia, defined as SpO2 <92% on room air, new receipt of supplemental oxygen to maintain SpO2 ≥92%, or increased supplemental oxygen to maintain SpO2 ≥92% for a patient on chronic oxygen therapy).
   4. sore throat
4. Laboratory-confirmed SARS-CoV-2 infection within the past 10 days prior to randomization.

Exclusion Criteria:

1. Prisoner
2. Pregnancy
3. Breast feeding
4. Symptoms of acute respiratory infection for >10 days before randomization
5. >48 hours between meeting inclusion criteria and randomization
6. Seizure disorder
7. Porphyria cutanea tarda
8. Diagnosis of Long QT syndrome
9. QTc >500 ms on electrocardiogram within 72 hours prior to enrollment
10. Known allergy to hydroxychloroquine, chloroquine, or amodiaquine
11. Receipt in the 12 hours prior to enrollment, or planned administration during the 5-day study period that treating clinicians feel cannot be substituted for another medication, of any of the following: amiodarone; cimetidine; dofetilide; phenobarbital; phenytoin; sotalol
12. Receipt of >1 dose of hydroxychloroquine or chloroquine in the 10 days prior to enrollment
13. Inability to receive enteral medications
14. Refusal or inability to be contacted on Day 15 for clinical outcome assessment if discharged prior to day 15
15. Previous enrollment in this trial
16. The treating clinical team does not believe equipoise exists regarding the use of hydroxychloroquine for the treatment of this patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 479 (Actual)
Dates: Start 2020-04-02 (Actual); Primary Completion 2020-06-19 (Actual); Study Completion 2020-07-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boyd Taylor Thompson, MD, Principal Investigator — Massachusetts General Hospital
Locations (40):
- United States (40):
  - University of Arizona, Tucson, Arizona
  - UCSF Fresno, Fresno, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - UC Davis Medical Center, Sacramento, California
  - UCSF Medical Center, San Francisco, California
  - Stanford University, Stanford, California
  - Medical Center of Aurora, Aurora, Colorado
  - University of Colorado Hospital, Aurora, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - University of Florida, Gainesville, Florida
  - University of Kentucky, Lexington, Kentucky
  - University Medical Center, New Orleans, Louisiana
  - Maine Medical Center, Portland, Maine
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - St. Vincent's Hospital, Worcester, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Henry Ford Medical Center, Detroit, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Montefiore Medical Center-Weiler, The Bronx, New York
  - Montefiore Medical Center-Moses, The Bronx, New York
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Wexner Medical Center, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - UPMC Presbyterian/Mercy/Shadyside, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Health Science Center, Houston, Texas
  - Intermountain Medical Center, Murray, Utah
  - University of Utah Hospital, Salt Lake City, Utah
  - VCU Medical Center, Richmond, Virginia
  - Harborview Medical Center, Seattle, Washington
  - Swedish Hospital First Hill, Seattle, Washington

REFERENCES:
- [Derived] Self WH, Semler MW, Leither LM, Casey JD, Angus DC, Brower RG, Chang SY, Collins SP, Eppensteiner JC, Filbin MR, Files DC, Gibbs KW, Ginde AA, Gong MN, Harrell FE Jr, Hayden DL, Hough CL, Johnson NJ, Khan A, Lindsell CJ, Matthay MA, Moss M, Park PK, Rice TW, Robinson BRH, Schoenfeld DA, Shapiro NI, Steingrub JS, Ulysse CA, Weissman A, Yealy DM, Thompson BT, Brown SM; National Heart, Lung, and Blood Institute PETAL Clinical Trials Network; Steingrub J, Smithline H, Tiru B, Tidswell M, Kozikowski L, Thornton-Thompson S, De Souza L, Hou P, Baron R, Massaro A, Aisiku I, Fredenburgh L, Seethala R, Johnsky L, Riker R, Seder D, May T, Baumann M, Eldridge A, Lord C, Shapiro N, Talmor D, O'Mara T, Kirk C, Harrison K, Kurt L, Schermerhorn M, Banner-Goodspeed V, Boyle K, Dubosh N, Filbin M, Hibbert K, Parry B, Lavin-Parsons K, Pulido N, Lilley B, Lodenstein C, Margolin J, Brait K, Jones A, Galbraith J, Peacock R, Nandi U, Wachs T, Matthay M, Liu K, Kangelaris K, Wang R, Calfee C, Yee K, Hendey G, Chang S, Lim G, Qadir N, Tam A, Beutler R, Levitt J, Wilson J, Rogers A, Vojnik R, Roque J, Albertson T, Chenoweth J, Adams J, Pearson S, Juarez M, Almasri E, Fayed M, Hughes A, Hillard S, Huebinger R, Wang H, Vidales E, Patel B, Ginde A, Moss M, Baduashvili A, McKeehan J, Finck L, Higgins C, Howell M, Douglas I, Haukoos J, Hiller T, Lyle C, Cupelo A, Caruso E, Camacho C, Gravitz S, Finigan J, Griesmer C, Park P, Hyzy R, Nelson K, McDonough K, Olbrich N, Williams M, Kapoor R, Nash J, Willig M, Ford H, Gardner-Gray J, Ramesh M, Moses M, Ng Gong M, Aboodi M, Asghar A, Amosu O, Torres M, Kaur S, Chen JT, Hope A, Lopez B, Rosales K, Young You J, Mosier J, Hypes C, Natt B, Borg B, Salvagio Campbell E, Hite RD, Hudock K, Cresie A, Alhasan F, Gomez-Arroyo J, Duggal A, Mehkri O, Hastings A, Sahoo D, Abi Fadel F, Gole S, Shaner V, Wimer A, Meli Y, King A, Terndrup T, Exline M, Pannu S, Robart E, Karow S, Hough C, Robinson B, Johnson N, Henning D, Campo M, Gundel S, Seghal S, Katsandres S, Dean S, Khan A, Krol O, Jouzestani M, Huynh P, Weissman A, Yealy D, Scholl D, Adams P, McVerry B, Huang D, Angus D, Schooler J, Moore S, Files C, Miller C, Gibbs K, LaRose M, Flores L, Koehler L, Morse C, Sanders J, Langford C, Nanney K, MdalaGausi M, Yeboah P, Morris P, Sturgill J, Seif S, Cassity E, Dhar S, de Wit M, Mason J, Goodwin A, Hall G, Grady A, Chamberlain A, Brown S, Bledsoe J, Leither L, Peltan I, Starr N, Fergus M, Aston V, Montgomery Q, Smith R, Merrill M, Brown K, Armbruster B, Harris E, Middleton E, Paine R, Johnson S, Barrios M, Eppensteiner J, Limkakeng A, McGowan L, Porter T, Bouffler A, Leahy JC, deBoisblanc B, Lammi M, Happel K, Lauto P, Self W, Casey J, Semler M, Collins S, Harrell F, Lindsell C, Rice T, Stubblefield W, Gray C, Johnson J, Roth M, Hays M, Torr D, Zakaria A, Schoenfeld D, Thompson T, Hayden D, Ringwood N, Oldmixon C, Ulysse C, Morse R, Muzikansky A, Fitzgerald L, Whitaker S, Lagakos A, Brower R, Reineck L, Aggarwal N, Bienstock K, Freemer M, Maclawiw M, Weinmann G, Morrison L, Gillespie M, Kryscio R, Brodie D, Zareba W, Rompalo A, Boeckh M, Parsons P, Christie J, Hall J, Horton N, Zoloth L, Dickert N, Diercks D. Effect of Hydroxychloroquine on Clinical Status at 14 Days in Hospitalized Patients With COVID-19: A Randomized Clinical Trial. JAMA. 2020 Dec 1;324(21):2165-2176. doi: 10.1001/jama.2020.22240. PMID 33165621
- [Derived] Casey JD, Johnson NJ, Semler MW, Collins SP, Aggarwal NR, Brower RG, Chang SY, Eppensteiner J, Filbin M, Gibbs KW, Ginde AA, Gong MN, Harrell F, Hayden DL, Hough CL, Khan A, Leither LM, Moss M, Oldmixon CF, Park PK, Reineck LA, Ringwood NJ, Robinson BRH, Schoenfeld DA, Shapiro NI, Steingrub JS, Torr DK, Weissman A, Lindsell CJ, Rice TW, Thompson BT, Brown SM, Self WH. Rationale and Design of ORCHID: A Randomized Placebo-controlled Clinical Trial of Hydroxychloroquine for Adults Hospitalized with COVID-19. Ann Am Thorac Soc. 2020 Sep;17(9):1144-1153. doi: 10.1513/AnnalsATS.202005-478SD. PMID 32492354
- See also: Website for the PETAL Network — http://petalnet.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Hydroxychloroquine: Participants assigned to the hydroxychloroquine arm will receive hydroxychloroquine sulfate 400 mg twice daily on the day of enrollment, then 200 mg twice daily for the next 4 days for a 5 day total course.
  Hydroxychloroquine: Hydroxychloroquine is available in 200 mg oral tablets of hydroxychloroquine sulfate.
  For this COVID-19 trial, we will use an oral or enteral dose of hydroxychloroquine 400 mg twice daily on the day of enrollment, then 200 mg twice daily for the next 4 days for a 5 day total course.
Period: Overall Study
Arm/Group | Hydroxychloroquine | Placebo
Started | 242 | 237
Completed | 242 | 237
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hydroxychloroquine | Placebo | Total
Number analyzed (Participants) | 242 | 237 | 479
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 58 [45 to 69] | 57 [43 to 68] | 57 [44 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107 | 105 | 212
  Male | 135 | 132 | 267
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: This measure was analyzed in participants with available data on race and ethnicity.
  Participants
    Non-Hispanic White: number analyzed (Participants) | 232 | 227 | 459
    Non-Hispanic White | 72 | 65 | 137
    Non-Hispanic Black: number analyzed (Participants) | 232 | 227 | 459
    Non-Hispanic Black | 57 | 55 | 112
    Hispanic: number analyzed (Participants) | 232 | 227 | 459
    Hispanic | 91 | 87 | 178
    Asian: number analyzed (Participants) | 232 | 227 | 459
    Asian | 4 | 7 | 11
    Native Hawaiian or other Pacific Islander: number analyzed (Participants) | 232 | 227 | 459
    Native Hawaiian or other Pacific Islander | 2 | 4 | 6
    Multi-race: number analyzed (Participants) | 232 | 227 | 459
    Multi-race | 1 | 1 | 2
    American Indian or Alaska Native: number analyzed (Participants) | 232 | 227 | 459
    American Indian or Alaska Native | 5 | 8 | 13
Living at home in the community prior to hospitalization [Count of Participants; unit: Participants] | 190 | 183 | 373
Body mass index [Median (Inter-Quartile Range); unit: kg/m^2] — Population: This measure was analyzed in participants with available data on body mass index
  kg/m^2
    number analyzed (Participants) | 226 | 219 | 445
    (all) | 31.3 [26.4 to 37.2] | 31.1 [27.2 to 36.5] | 31.1 [26.9 to 36.9]
Chronic Conditions [Count of Participants; unit: Participants]
  Hypertension | 136 | 117 | 253
  Diabetes | 88 | 78 | 166
  Chronic kidney disease | 28 | 14 | 42
  Chronic artery disease | 19 | 23 | 42
  Chronic obstructive pulmonary disease | 18 | 21 | 39
Location at time of randomization [Count of Participants; unit: Participants] — Population: Measure was analyzed in participants with available data on location at time of randomization.
  Participants
    Hospital ward: number analyzed (Participants) | 228 | 224 | 452
    Hospital ward | 157 | 132 | 289
    Intensive care unit: number analyzed (Participants) | 228 | 224 | 452
    Intensive care unit | 37 | 54 | 91
    Emergency department: number analyzed (Participants) | 228 | 224 | 452
    Emergency department | 34 | 38 | 72
Symptoms of acute respiratory infection [Count of Participants; unit: Participants]
  Shortness of breath | 175 | 168 | 343
  Cough | 143 | 140 | 283
  Fever (temperature > 37.5 degrees celsius) | 138 | 132 | 270
Duration of symptoms prior to randomization [Median (Inter-Quartile Range); unit: days] | 5 [3 to 7] | 5 [3 to 7] | 5 [3 to 7]
Time between hospital presentation and randomization [Median (Inter-Quartile Range); unit: hours] — Defined as the time of the first contact with an acute care hospital during the health care episode that resulted in the hospitalization during which the patient was enrolled. For patients who initially presented to the emergency department, time of hospital presentation was the time of emergency department arrival. For patients directly hospitalized without presenting to the emergency department, time of hospital presentation was the time of arrival at the admission unit. Population: Measure was analyzed in participants who had available data for date of hospital presentation.
  hours
    number analyzed (Participants) | 240 | 234 | 474
    (all) | 22.2 [14.6 to 33.1] | 22.7 [14.1 to 29.9] | 22.5 [14.3 to 31.6]
COVID outcomes scale category at randomization [Count of Participants; unit: Participants] — The COVID Outcomes Scale is a 7-category ordinal scale that classifies a patient's clinical status. Lower scores indicate more severely ill clinical status. Patients in the following categories at baseline were not eligible for enrollment: category 1 (death); category 6 (not hospitalized and unable to perform normal activities); and category 7 (not hospitalized and able to perform normal activities).
  Participants
    2: Hospitalized, receiving ECMO or invasive mechanical ventilation | 13 | 19 | 32
    3: Hospitalized, receiving noninvasive ventilation or nasal high flow oxygen | 28 | 27 | 55
    4: Hospitalized, receiving supplemental oxygen without positive pressure or high flow | 116 | 108 | 224
    5: Hospitalized, not receiving supplemental oxygen | 85 | 83 | 168
Vasopressor use at enrollment [Count of Participants; unit: Participants] | 8 | 20 | 28
Total SOFA score at enrollment [Median (Inter-Quartile Range); unit: score] — The SOFA score categorizes illness severity based on organ dysfunction across 6 organ systems: respiratory, coagulation, liver, cardiovascular, central nervous system, and kidney. SOFA scores range from 0 to 24, with higher scores indicating greater illness severity. A SOFA score of 2 indicates moderate dysfunction in 1 organ system or mild dysfunction in 2 organ systems.
  score | 2 [1 to 4] | 2 [1 to 4] | 2 [1 to 4]
White blood cell count [Median (Inter-Quartile Range); unit: cells ×10^3/μL] — Normal range for WBC: 3.9-10.7 Population: Measure is analyzed in participants with available data on white blood cell count.
  cells ×10^3/μL
    number analyzed (Participants) | 224 | 218 | 442
    (all) | 6.0 [4.3 to 7.9] | 5.9 [4.1 to 7.7] | 5.9 [4.2 to 7.8]
Platelet count [Median (Inter-Quartile Range); unit: cells ×10^3/μL] — Normal range for platelet: 135-371 Laboratory normal ranges were reported base on the clinical laboratory normal ranges from Vanderbilt University Medical Center. Normal ranges may vary across laboratories. Population: Measure is analyzed in participants with available data on platelet count.
  cells ×10^3/μL
    number analyzed (Participants) | 237 | 230 | 467
    (all) | 199 [151 to 247] | 200 [147 to 251] | 199 [148 to 250]
Creatinine [Median (Inter-Quartile Range); unit: mg/dL] — Normal range for creatinine: 0.57-1.11 Laboratory normal ranges were reported base on the clinical laboratory normal ranges from Vanderbilt University Medical Center. Normal ranges may vary across laboratories. Population: Measure was analyzed in participants with available data on creatinine.
  mg/dL
    number analyzed (Participants) | 235 | 231 | 466
    (all) | 0.95 [0.75 to 1.47] | 0.90 [0.75 to 1.25] | 0.91 [0.75 to 1.36]
Aspartate aminotransferase [Median (Inter-Quartile Range); unit: U/L] — Normal range for aspartate aminotransferase: 5-40 Laboratory normal ranges were reported base on the clinical laboratory normal ranges from Vanderbilt University Medical Center. Normal ranges may vary across laboratories. Population: Measure is analyzed in participants with available data on aspartate aminotransferase.
  U/L
    number analyzed (Participants) | 173 | 184 | 357
    (all) | 39 [29 to 62] | 45 [31 to 70] | 41 [29 to 66]
Alanine aminotransferase [Median (Inter-Quartile Range); unit: U/L] — Normal range for alanine aminotransferase: 0-55 Laboratory normal ranges were reported base on the clinical laboratory normal ranges from Vanderbilt University Medical Center. Normal ranges may vary across laboratories. Population: Measure was analyzed in participants with available data on alanine aminotransferase.
  U/L
    number analyzed (Participants) | 174 | 183 | 357
    (all) | 30 [18 to 47] | 34 [23 to 62] | 31 [20 to 56]
Bilateral infiltrates on chest imaging [Count of Participants; unit: Participants] — Reported chest imaging interpretations were based on final interpretation from radiologists. Population: This measure was analyzed in participants with available data on bilateral infiltrates on chest imaging.
  Participants
    number analyzed (Participants) | 230 | 230 | 460
    (all) | 147 | 145 | 292
QTc interval [Median (Inter-Quartile Range); unit: milliseconds] — Reported QTc was based on automated readings. Population: This measure was analyzed in participants with available data on QTc interval.
  milliseconds
    number analyzed (Participants) | 242 | 236 | 478
    (all) | 430 [414 to 452] | 435 [416 to 452] | 433 [415 to 452]

OUTCOME MEASURES:

1. Primary Outcome: COVID Outcomes Scale Score on Study Day 15 (14 Days After Randomization)
Description: We will determine the COVID Ordinal Scale for all patients on study day 15
  COVID Ordinal Scale defined as:
  1. Death
  2. Hospitalized on invasive mechanical ventilation or ECMO ( extracorporeal membrane oxygenation)
  3. Hospitalized on non-invasive ventilation or high flow nasal cannula
  4. Hospitalized on supplemental oxygen
  5. Hospitalized not on supplemental oxygen
  6. Not hospitalized with limitation in activity (continued symptoms)
  7. Not hospitalized without limitation in activity (no symptoms)
Time Frame: Assessed on study day 15
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 242 | 237
score on a scale | 6 [4 to 7] | 6 [4 to 7]
Statistical Analysis 1: Comparison: Hydroxychloroquine vs Placebo; Outcome measure was adjusted for age, sex, baseline COVID Outcome Scale category, baseline Sequential Organ Failure Assessment score, and duration of acute respiratory infection symptoms prior to randomization; Test type: Superiority; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.73 to 1.42] — Odds ratios greater than 1.0 indicated more favorable outcomes for patients in the hydroxychloroquine group compared with the placebo group

2. Secondary Outcome: COVID Ordinal Outcomes Scale on Study Day 3 (2 Days After Randomization)
Description: We will determine the COVID Ordinal Scale for all patients on study day 3
  COVID Ordinal Scale defined as:
  1. Death
  2. Hospitalized on invasive mechanical ventilation or ECMO ( extracorporeal membrane oxygenation)
  3. Hospitalized on non-invasive ventilation or high flow nasal cannula
  4. Hospitalized on supplemental oxygen
  5. Hospitalized not on supplemental oxygen
  6. Not hospitalized with limitation in activity (continued symptoms)
  7. Not hospitalized without limitation in activity (no symptoms)
Time Frame: assessed on study day 3
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 242 | 237
score on a scale | 4 [3 to 5] | 4 [3 to 5]
Statistical Analysis 1: Comparison: Hydroxychloroquine vs Placebo; Outcome measure was adjusted for: age, sex, baseline COVID Outcome Scale category, baseline Sequential Organ Failure Assessment score, and duration of acute respiratory infection symptoms prior to randomization; Test type: Superiority; Odds Ratio (OR) = 1.28, 95% CI 2-sided [0.90 to 1.81] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: COVID Ordinal Outcomes Scale on Study Day 8 (7 Days After Randomization)
Description: We will determine the COVID Ordinal Scale on study day 8
  COVID Ordinal Scale defined as:
  1. Death
  2. Hospitalized on invasive mechanical ventilation or ECMO ( extracorporeal membrane oxygenation)
  3. Hospitalized on non-invasive ventilation or high flow nasal cannula
  4. Hospitalized on supplemental oxygen
  5. Hospitalized not on supplemental oxygen
  6. Not hospitalized with limitation in activity (continued symptoms)
  7. Not hospitalized without limitation in activity (no symptoms)
Time Frame: assessed on study day 8
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 242 | 237
score on a scale | 5 [4 to 7] | 6 [3 to 6]
Statistical Analysis 1: Comparison: Hydroxychloroquine vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Odds Ratio (OR) = 1.16, 95% CI 2-sided [0.84 to 1.61] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: COVID Ordinal Outcomes Scale on Study Day 29 (28 Days After Randomization)
Description: We will determine the COVID Ordinal Scale on study day 29
  COVID Ordinal Scale defined as:
  1. Death
  2. Hospitalized on invasive mechanical ventilation or ECMO ( extracorporeal membrane oxygenation)
  3. Hospitalized on non-invasive ventilation or high flow nasal cannula
  4. Hospitalized on supplemental oxygen
  5. Hospitalized not on supplemental oxygen
  6. Not hospitalized with limitation in activity (continued symptoms)
  7. Not hospitalized without limitation in activity (no symptoms)
Time Frame: assessed on study day 29
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 242 | 237
score on a scale | 6 [6 to 7] | 6 [6 to 7]
Statistical Analysis 1: Comparison: Hydroxychloroquine vs Placebo; Outcome measure is adjusted for : age, sex, baseline COVID Outcome Scale category, baseline Sequential Organ Failure Assessment score, and duration of acute respiratory infection symptoms prior to randomization; Test type: Superiority; Odds Ratio (OR) = 0.97, 95% CI 2-sided [0.69 to 1.38] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: All-location, All-cause Mortality Assessed on Study Day 15 (14 Days After Randomization)
Description: Vital status of the patient on day 15 will be determined using any of the following methods: medical record review, phone calls to patient or proxy.
  There were two patients for whom we were unable to collect their vital status.
Time Frame: assessed on study day 15
Population: Outcome was measured in participants with available data on vital status. One patient in the hydroxychloroquine group and one patient in the placebo group were lost to follow-up for vital status.
Measure: Count of Participants; unit: Participants
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 241 | 236
Participants | 18 | 14
Statistical Analysis 1: Comparison: Hydroxychloroquine vs Placebo; Test type: Superiority; Odds Ratio (OR) = 1.56, 95% CI 2-sided [0.68 to 3.57] — Odds ratios greater than 1.0 indicated less favorable outcomes for patients in the hydroxychloroquine group compared with the placebo group

6. Secondary Outcome: All-location, All-cause Mortality Assessed on Study Day 29 (28 Days After Randomization)
Description: Vital status of the patient at day 28 will be determined using any of the following methods: medical record review, phone calls to patient or proxy.
  There were two patients for whom we were unable to collect their vital status.
Time Frame: assessed on study day 29
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 241 | 236
Participants | 25 | 25
Statistical Analysis 1: Comparison: Hydroxychloroquine vs Placebo; Test type: Superiority; Odds Ratio (OR) = 1.07, 95% CI 2-sided [0.54 to 2.09] — [estimate comment as in outcome 5, analysis 1]

7. Secondary Outcome: Number of Patients Dead or With Receipt of ECMO Between Enrollment and Day 28
Description: We will determine the number of patients who are either dead or on ECMO ( extracorporeal membrane oxygenation) between enrollment and day 28
Time Frame: Enrollment to Day 28
Population: Outcome was measured in participants with available data on vital status or ECMO. One patient in the hydroxychloroquine group and one patient in the placebo group were lost to follow-up for vital status.
Measure: Count of Participants; unit: Participants
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 241 | 236
Participants | 29 | 28
Statistical Analysis 1: Comparison: Hydroxychloroquine vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Odds Ratio (OR) = 1.13, 95% CI 2-sided [0.60 to 2.14] — [estimate comment as in outcome 5, analysis 1]

8. Secondary Outcome: Oxygen-free Days Through Day 28
Description: The number of calendar days between randomization and 28 days later that the patient is alive and without the use of oxygen therapy. Patients who die prior to day 28 are assigned zero oxygen free days.
Time Frame: 28 days after randomization
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 242 | 237
days | 21 [0 to 27] | 20 [0 to 27]
Statistical Analysis 1: Comparison: Hydroxychloroquine vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Odds Ratio (OR) = 0.96, 95% CI 2-sided [0.68 to 1.34] — [estimate comment as in outcome 1, analysis 1]

9. Secondary Outcome: Ventilator-free Days Through Day 28
Description: Ventilator-free days is defined to be 28 days minus the duration of mechanical ventilation through day 28. Participants who do not survive to day 28 are assigned zero ventilator-free days.
Time Frame: 28 days after randomization
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 242 | 237
days | 28 [28 to 28] | 28 [28 to 28]
Statistical Analysis 1: Comparison: Hydroxychloroquine vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Odds Ratio (OR) = 1.26, 95% CI 2-sided [0.76 to 2.08] — [estimate comment as in outcome 1, analysis 1]

10. Secondary Outcome: Vasopressor-free Days Through Day 28
Description: The number of calendar days between randomization and 28 days later that the patient is alive and without the use of vasopressor therapy. Patients who die prior to day 28 are assigned zero vasopressor free days.
Time Frame: 28 days after randomization
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 242 | 237
days | 28 [28 to 28] | 28 [28 to 28]
Statistical Analysis 1: Comparison: Hydroxychloroquine vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Odds Ratio (OR) = 1.03, 95% CI 2-sided [0.61 to 1.72] — [estimate comment as in outcome 1, analysis 1]

11. Secondary Outcome: ICU-free Days to Day 28
Description: The number of days spent out of the ICU to day 28. Patients who die prior to day 28 are assigned zero ICU free days.
Time Frame: 28 days after randomization
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 242 | 237
days | 28 [21 to 28] | 28 [18 to 28]
Statistical Analysis 1: Comparison: Hydroxychloroquine vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Odds Ratio (OR) = 1.26, 95% CI 2-sided [0.84 to 1.88] — [estimate comment as in outcome 1, analysis 1]

12. Secondary Outcome: Hospital-free Days to Day 28
Description: Defined as 28 days minus the number of days from randomization to discharge home.If a patient has not been discharged home prior to day 28 or dies prior to day 28, hospital free days will be zero.
Time Frame: 28 days after randomization
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 242 | 237
days | 21 [11 to 24] | 20 [10 to 24]
Statistical Analysis 1: Comparison: Hydroxychloroquine vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Odds Ratio (OR) = 1.17, 95% CI 2-sided [0.85 to 1.61] — [estimate comment as in outcome 1, analysis 1]

13. Other Pre Specified Outcome: Number of Patients With Seizures to Day 28
Description: We will determine the number of patients that experience seizure between randomization and day 28
Time Frame: 28 days after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 242 | 237
Participants | 1 | 0
Statistical Analysis 1: Comparison: Hydroxychloroquine vs Placebo; Test type: Superiority; Risk Difference (RD) = 0.4, 95% CI 2-sided [-1.0 to 1.8]

14. Other Pre Specified Outcome: Number of Patients With Atrial Arrhythmia to Day 28
Description: We will determine the number of patients that experience atrial arrhythmia between randomization and day 28
Time Frame: 28 days after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 242 | 237
Participants | 15 | 11
Statistical Analysis 1: Comparison: Hydroxychloroquine vs Placebo; Test type: Superiority; Odds Ratio (OR) = 1.36, 95% CI 2-sided [0.61 to 3.02] — [estimate comment as in outcome 5, analysis 1]

15. Other Pre Specified Outcome: Number of Patients With Ventricular Arrhythmia to Day 28
Description: We will determine the number of patients that experience ventricular arrhythmia between randomization and day 28
Time Frame: 28 days after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 242 | 237
Participants | 5 | 6
Statistical Analysis 1: Comparison: Hydroxychloroquine vs Placebo; Test type: Superiority; Odds Ratio (OR) = 0.81, 95% CI 2-sided [0.24 to 2.70] — [estimate comment as in outcome 5, analysis 1]

16. Other Pre Specified Outcome: Number of Patients With Cardiac Arrest to Day 28
Description: We will determine the number of patients that experience cardiac arrest between randomization and day 28
Time Frame: 28 days after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 242 | 237
Participants | 10 | 4
Statistical Analysis 1: Comparison: Hydroxychloroquine vs Placebo; Test type: Superiority; Odds Ratio (OR) = 2.51, 95% CI 2-sided [0.78 to 8.12] — [estimate comment as in outcome 5, analysis 1]

17. Other Pre Specified Outcome: Number of Patients With Elevation in Aspartate Aminotransferase or Alanine Aminotransferase to Twice the Local Upper Limit of Normal to Day 28
Description: We will determine the number of patients that experience elevation in aspartate aminotransferase or alanine aminotransferase to twice the local upper limit of normal between randomization and day 28
Time Frame: 28 days after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 242 | 237
Participants | 50 | 65
Statistical Analysis 1: Comparison: Hydroxychloroquine vs Placebo; Test type: Superiority; Odds Ratio (OR) = 0.69, 95% CI 2-sided [0.45 to 1.05] — [estimate comment as in outcome 5, analysis 1]

18. Other Pre Specified Outcome: Number of Patients With Acute Pancreatitis Arrest to Day 28
Description: We will determine the number of patients that experience acute pancreatitis between randomization and day 28
Time Frame: 28 days after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 242 | 237
Participants | 5 | 6
Statistical Analysis 1: Comparison: Hydroxychloroquine vs Placebo; Test type: Superiority; Odds Ratio (OR) = 0.81, 95% CI 2-sided [0.24 to 2.70] — [estimate comment as in outcome 5, analysis 1]

19. Other Pre Specified Outcome: Number of Patients With Acute Kidney Injury to day28
Description: We will determine the number of patients that experience acute kidney injury between randomization and day 28
Time Frame: 28 days after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 242 | 237
Participants | 37 | 37
Statistical Analysis 1: Comparison: Hydroxychloroquine vs Placebo; Test type: Superiority; Odds Ratio (OR) = 0.97, 95% CI 2-sided [0.59 to 1.59] — [estimate comment as in outcome 5, analysis 1]

20. Other Pre Specified Outcome: Number of Patients With Receipt of Renal Replacement Therapy to Day 28
Description: We will determine the number of patients that experience renal replacement therapy between randomization and day 28
Time Frame: 28 days after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 242 | 237
Participants | 10 | 14
Statistical Analysis 1: Comparison: Hydroxychloroquine vs Placebo; Test type: Superiority; Odds Ratio (OR) = 0.69, 95% CI 2-sided [0.30 to 1.58] — [estimate comment as in outcome 5, analysis 1]

21. Other Pre Specified Outcome: Number of Patients With Symptomatic Hypoglycemia to Day 28
Description: We will determine the number of patients that experience symptomatic hypoglycemia between randomization and day 28
Time Frame: 28 days after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 242 | 237
Participants | 10 | 8
Statistical Analysis 1: Comparison: Hydroxychloroquine vs Placebo; Test type: Superiority; Odds Ratio (OR) = 1.23, 95% CI 2-sided [0.48 to 3.18] — [estimate comment as in outcome 5, analysis 1]

22. Other Pre Specified Outcome: Number of Patients With Neutropenia to Day 28
Description: We will determine the number of patients that experience neutropenia between randomization and day 28
Time Frame: 28 days after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 242 | 237
Participants | 4 | 4
Statistical Analysis 1: Comparison: Hydroxychloroquine vs Placebo; Test type: Superiority; Odds Ratio (OR) = 0.98, 95% CI 2-sided [0.24 to 3.96] — [estimate comment as in outcome 5, analysis 1]

23. Other Pre Specified Outcome: Number of Patients With Lymphopenia to Day 28
Description: We will determine the number of patients that experience lymphopenia between randomization and day 28
Time Frame: 28 days after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 242 | 237
Participants | 92 | 87
Statistical Analysis 1: Comparison: Hydroxychloroquine vs Placebo; Test type: Superiority; Odds Ratio (OR) = 1.06, 95% CI 2-sided [0.73 to 1.53] — [estimate comment as in outcome 5, analysis 1]

24. Other Pre Specified Outcome: Number of Patients With Anemia to Day 28
Description: We will determine the number of patients that experience anemia between randomization and day 28
Time Frame: 28 days after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 242 | 237
Participants | 139 | 120
Statistical Analysis 1: Comparison: Hydroxychloroquine vs Placebo; Test type: Superiority; Odds Ratio (OR) = 1.32, 95% CI 2-sided [0.92 to 1.89] — [estimate comment as in outcome 5, analysis 1]

25. Other Pre Specified Outcome: Number of Patients With Thrombocytopenia to Day 28
Description: We will determine the number of patients that experience thrombocytopenia between randomization and day 28
Time Frame: 28 days after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 242 | 237
Participants | 4 | 5
Statistical Analysis 1: Comparison: Hydroxychloroquine vs Placebo; Test type: Superiority; Odds Ratio (OR) = 0.78, 95% CI 2-sided [0.21 to 2.94] — [estimate comment as in outcome 5, analysis 1]

26. Other Pre Specified Outcome: Number of Patients With Severe Dermatologic Reaction to Day 28
Description: We will determine the number of patients that experience severe dermatologic reaction between randomization and day 28
Time Frame: 28 days after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 242 | 237
Participants | 1 | 1
Statistical Analysis 1: Comparison: Hydroxychloroquine vs Placebo; Test type: Superiority; Odds Ratio (OR) = 0.98, 95% CI 2-sided [0.06 to 15.74] — [estimate comment as in outcome 5, analysis 1]

27. Other Pre Specified Outcome: Time to Recovery, Defined as Time to Reaching Level 5, 6, or 7 on the COVID Outcomes Scale, Which is the Time to the Earlier of Final Liberation From Supplemental Oxygen or Hospital Discharge
Description: Time to recovery, defined as time to reaching level 5, 6, or 7 on the COVID Outcomes Scale, which is the time to the earlier of final liberation from supplemental oxygen or hospital discharge. Patients who die prior to day 28 are assigned 28 days for time to recovery.
Time Frame: 28 days after randomization
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 242 | 237
days | 5 [1 to 14] | 6 [1 to 15]
Statistical Analysis 1: Comparison: Hydroxychloroquine vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Odds Ratio (OR) = 0.97, 95% CI 2-sided [0.69 to 1.35] — [estimate comment as in outcome 5, analysis 1]

ADVERSE EVENTS:
Time Frame: Subjects were assessed for adverse events from enrollment through study day 29 or discharge, whichever occurs first. Investigators will determine if the event is serious or related to study drug.
Groups:
- Hydroxychlorquine: Participants assigned to the hydroxychloroquine arm will receive hydroxychloroquine sulfate 400 mg twice daily on the day of enrollment, then 200 mg twice daily for the next 4 days for a 5 day total course.
  Hydroxychloroquine: Hydroxychloroquine is available in 200 mg oral tablets of hydroxychloroquine sulfate.
  For this COVID-19 trial, we will use an oral or enteral dose of hydroxychloroquine 400 mg twice daily on the day of enrollment, then 200 mg twice daily for the next 4 days for a 5 day total course.
Arm/Group | Hydroxychlorquine | Placebo
All-Cause Mortality (participants affected / at risk) | 25/242 | 25/237
Serious Adverse Events (participants affected / at risk) | 14/242 | 11/237
Other Adverse Events (participants affected / at risk) | 30/242 | 21/237
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydroxychlorquine (N=242) | Placebo (N=237)
Cardiac Arrest (Cardiac disorders) | 0 (0) | 2 (2)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal Distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bleeding Gastrointestinal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gall stones (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea, Vomiting, Hematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Obstruction Bowel (Gastrointestinal disorders) | 1 (1) | 0 (0)
Death (General disorders) | 2 (2) | 0 (0)
Hypokalemia (Investigations) | 0 (0) | 1 (1)
Reaction Nonspecific (Investigations) | 1 (1) | 1 (1)
Hematoma Muscle (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Edema Cerebral (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Stroke (Nervous system disorders) | 1 (1) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hemorrhage Retroperitoneal (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydroxychlorquine (N=242) | Placebo (N=237)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial Arrythmia (Cardiac disorders) | 1 (1) | 2 (2)
Bradycardia (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Chest Pain (Cardiac disorders) | 2 (2) | 0 (0)
Conduction Disorder (Cardiac disorders) | 0 (0) | 1 (1)
EKG Abnormality: Non-Specific (Cardiac disorders) | 0 (0) | 1 (1)
Premature Ventricular Contractions (Cardiac disorders) | 1 (1) | 1 (1)
Prolonged QTc (Cardiac disorders) | 2 (2) | 3 (3)
Sinus Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Hypoglycemia (Endocrine disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Nausea, Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea, Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Contrast Extravasation (General disorders) | 1 (1) | 0 (0)
Allergic Reaction (Immune system disorders) | 1 (1) | 0 (0)
ALT Increased (Investigations) | 1 (1) | 0 (0)
AST Increased (Investigations) | 1 (1) | 0 (0)
Multiple Liver Function Tests Abnormal (Investigations) | 10 (10) | 3 (3)
Headache (Nervous system disorders) | 3 (3) | 2 (2)
Neuropathy Peripheral (Nervous system disorders) | 0 (0) | 1 (1)
Kidney Function Abnormal (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Itching (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 1 (1)
Vagal Reaction (Vascular disorders) | 1 (1) | 0 (0)
Nosebleed (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2020-06-04): https://cdn.clinicaltrials.gov/large-docs/91/NCT04332991/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-17): https://cdn.clinicaltrials.gov/large-docs/91/NCT04332991/SAP_001.pdf